CLINICAL TRIAL: NCT01154426
Title: Phase I Study of ABT-888 in Combination With Gemcitabine in Patients With Advanced Malignancies
Brief Title: ABT-888 and Gemcitabine Hydrochloride in Treating Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2011-01473; NCI-2011-01473 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000673613; 09-012 (Other: University of Pittsburgh Cancer Institute (UPCI)); 8324 (Other: CTEP); P30CA047904 (NIH); U01CA099168 (NIH)
Record Dates: First submitted 2010-06-29; First posted 2010-06-30 (Estimated); Last update posted 2015-07-02 (Estimated); Status verified 2014-12

CONDITIONS: Adult Solid Neoplasm; BRCA1 Mutation Carrier; BRCA2 Mutation Carrier
MeSH Terms: interventions — Gemcitabine; veliparib

ARMS (1):
- Treatment (gemcitabine hydrochloride and ABT-888) (Experimental): Patients receive oral ABT-888 twice daily on days 1-14 and gemcitabine hydrochloride IV over 30 minutes on days 1, 8, and 15. Courses repeat every 21* days in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: Diagnostic Laboratory Biomarker Analysis; Drug: Gemcitabine Hydrochloride; Other: Pharmacological Study; Drug: Veliparib

INTERVENTIONS:
Other: Diagnostic Laboratory Biomarker Analysis — Correlative studies
Drug: Gemcitabine Hydrochloride — Given IV
  Other Names: dFdCyd; Difluorodeoxycytidine Hydrochloride; Gemzar; LY-188011
Other: Pharmacological Study — Correlative studies
Drug: Veliparib — Given orally
  Other Names: ABT-888; PARP-1 inhibitor ABT-888

SUMMARY:
This phase I trial is studying the side effects and best dose of giving ABT-888 together with gemcitabine hydrochloride in treating patients with advanced solid tumors. ABT-888 may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Drugs used in chemotherapy, such as gemcitabine hydrochloride, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving ABT-888 together with gemcitabine hydrochloride may kill more tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Establish the maximum-tolerated dose (MTD) and dose-limiting toxicities (DLTs) of the combination of ABT-888 and gemcitabine (gemcitabine hydrochloride) in patients with advanced solid tumors.

SECONDARY OBJECTIVES:

I. Establish the safety and tolerability of the combination of ABT-888 and gemcitabine in patients with solid tumors.

II. Determine the effects of ABT-888 and gemcitabine treatment on DNA damage response by analysis of markers such as Ataxia telangiectasia mutated (ATM) in peripheral blood mononuclear cells (PBMCs).

III. Determine the pharmacokinetics of ABT-888 and gemcitabine when administered in combination.

IV. Determine the generation of gemcitabine triphosphate in PBMCs. V. Document any evidence of antitumor response.

OUTLINE: This is a dose-escalation study.

Patients receive oral ABT-888 twice daily on days 1-14 and gemcitabine hydrochloride IV over 30 minutes on days 1, 8, and 15. Courses repeat every 21* days in the absence of disease progression or unacceptable toxicity.

After completion of study therapy, patients are followed up for at least 4 weeks.

NOTE: *Patients previously enrolled on a 4-week schedule (ABT-888 twice daily on days 1-21 with gemcitabine IV over 30 minutes once weekly on days 1, 8, and 15, and courses repeating every 28 days) will continue on the 4-week schedule.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed solid tumors meeting 1 of the following criteria:

  * Progressive disease following standard therapy
  * Disease for which acceptable standard treatment options do not exist
* May have received 0-2 prior chemotherapeutic regimens (single-agent or combination chemotherapies)
* Willing to undergo BRCA mutation analysis

  * Known BRCA mutations allowed
  * All patients, at any dose level, without a known BRCA mutation undergo screening with the BRCAPRO program to assess the likelihood of having a BRCA mutation
  * Patients with a BRCAPRO likelihood of gene mutation of ≥ 20% must undergo BRCA gene testing by the Myriad Genetic Laboratories in order to participate in the study

    * Patients are eligible whether they have a known deleterious BRCA 1 or 2 mutation or a mutation of uncertain significance
* No CNS disease (e.g., brain metastases or glioma)
* No active seizure or history of seizure disorder
* ECOG performance status 0-2 (Karnofsky 60-100%)
* Life expectancy > 3 months
* ANC ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* Bilirubin < 2.0 mg/dL
* AST and ALT < 3 times upper limit of normal
* Creatinine normal OR creatinine clearance > 50 mL/min
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* Able to swallow pills
* HIV-positive patients allowed provided that CD4 counts are < 500 and not on protease inhibitors
* No uncontrolled diarrhea
* No uncontrolled intercurrent illness including, but not limited to, any of the following:

  * Ongoing or active infection
  * Symptomatic congestive heart failure
  * Unstable angina pectoris
  * Cardiac arrhythmia
  * Psychiatric illness or social situations that would limit compliance with study requirements
* No other concurrent anticancer therapies or agents
* More than 4 weeks since prior major surgery, radiotherapy, or chemotherapy (6 weeks for mitomycin C or nitrosoureas) and recovered
* Prior gemcitabine hydrochloride or PARP inhibition therapy, including ABT-888, allowed

  * No prior combination of gemcitabine hydrochloride and any PARP inhibitor
* Concurrent bisphosphonate IV allowed provided treatment was initiated before study therapy (for patients with bone metastases or hypercalcemia)
* Patients with prostate cancer must continue luteinizing-hormone releasing-hormone agonist therapy and discontinue antiandrogens (≥ 6 weeks since bicalutamide and ≥ 4 weeks since flutamide)
* No other concurrent investigational agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2010-05; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
MTD of ABT-888 and gemcitabine hydrochloride, determined according to incidence of DLT graded using the NCI CTCAE version 4.0 | 3 weeks

SECONDARY OUTCOMES:
Adverse events as assessed by NCI CTCAE v 4.0 | Up to 4 weeks after completion of study treatment
  The maximum grade of toxicity for each category of interest will be recorded for each patient and the summary results will be tabulated by category and grade. We will describe all DLTs and other serious (≥ grade 3) on a patient-by-patient basis; descriptions will include dose level and any relevant baseline data. Statistics on the number of cycles received by patients and any dose reductions will be tabulated.
Plasma concentrations of gemcitabine hydrochloride and ABT-888 | Pre-drug, 25, 60, and 90 min, 2, 3, 4, 6, and 8 hours post-ABT-888 on day -2; pre-drug, 15, 25 (before end of gemcitabine infusion), 60, and 90 min, 2, 3, 4, 6, 8, 24, and 48 h after the start of gemcitabine hydrochloride infusion on day 1 of course 1
  Plasma concentration versus time data will be analyzed non-compartmentally using PK Solutions 2.0. Data may also be analyzed using compartmental methods as implemented by the ADAPT computer program or a suitable commercially available software package. Relationships between pharmacokinetic and pharmacodynamic data will be explored and evaluated using the ADAPT computer program or a suitable commercially available software packages.
Response (complete or partial response) | Up to 4 weeks after completion of study treatment
  Responses and incidence of stable disease will be tabulated by disease diagnosis and by dose level; no formal statistical analyses are planned.

CONTACTS AND LOCATIONS:
Overall Officials: Ronald Stoller, Principal Investigator — University of Pittsburgh Cancer Institute (UPCI)
Locations (4):
- United States (4):
  - Penn State Milton S Hershey Medical Center, Hershey, Pennsylvania
  - UPMC-Magee Womens Hospital, Pittsburgh, Pennsylvania
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania
  - University of Pittsburgh Cancer Institute, Pittsburgh, Pennsylvania

REFERENCES:
- [Derived] Manzo J, Puhalla S, Pahuja S, Ding F, Lin Y, Appleman L, Tawbi H, Stoller R, Lee JJ, Diergaarde B, Kiesel BF, Yu J, Tan AR, Belani CP, Chew H, Garcia AA, Morgan RJ, Wahner Hendrickson AE, Visscher DW, Hurley RM, Kaufmann SH, Swisher EM, Oesterreich S, Katz T, Ji J, Zhang Y, Parchment RE, Chen A, Duan W, Giranda V, Shepherd SP, Ivy SP, Chu E, Beumer JH; ETCTN-8282 study team. A phase 1 and pharmacodynamic study of chronically-dosed, single-agent veliparib (ABT-888) in patients with BRCA1- or BRCA2-mutated cancer or platinum-refractory ovarian or triple-negative breast cancer. Cancer Chemother Pharmacol. 2022 May;89(5):721-735. doi: 10.1007/s00280-022-04430-6. Epub 2022 Apr 18. PMID 35435472